CLINICAL TRIAL: NCT00563420
Title: Early Lung Cancer Detection in Patients With Sputum Cytology and Autofluorescence Bronchoscopy in People at High Risk of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Non-Randomized | Purpose: Diagnostic
Other Study IDs: EC 1621-01; HARECCTR0500035
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Lung Neoplasms
Keywords: Lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy

SUMMARY:
Lung cancer is the commonest malignant disease with a 5-year survival of 14%. In Hong Kong, it accounts for about 30% of all cancer death. The poor prognosis of lung cancer is due largely to the late clinical presentation of the disease. In order to improve the prognosis of lung cancer, an obvious approach is to develop sensitive methods for detecting lung cancer at much earlier stages when treatment is more likely to be curative.

However, the best way for identifying early lung cancer is still need to be determined. We hypothesis that by examining specimens that contain shed bronchial epithelial cells i.e. sputum, lung cancer can be sampled in its earliest possible phase. And by using autofluorescence bronchoscopy, a system specifically designed to detect early lung cancer/pre-invasive lesions, to identify the source of abnormal cells, we may able to detect eraly lung cancer and followed by curative treatment to improve the prognosis of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Current or ex-smokers who have smoked at least 20-pack-years (e.g. 1 pack per day for 20 years or more)
* Informed consent

Exclusion Criteria:

* Known malignant disease
* Unstable major medical disease
* Bleeding disorder
* Unwilling to have a bronchoscopy
* Women currently pregnant or nursing
* Known reaction to xylocaine, a local anaesthesia agent used for bronchoscopy

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Number of early stage lung cancer/precancerous lesion detected | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Bing Lam, Dr, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China